CLINICAL TRIAL: NCT03487172
Title: A Randomized, Split-body Clinical Trial of Poly-L-lactic Acid (Sculptra Aesthetic) for the Treatment of Upper Knee Skin Laxity
Brief Title: Sculptra Aesthetic for the Treatment of Upper Knee Skin Laxity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sculptra Knees
Record Dates: First submitted 2018-03-16; First posted 2018-04-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Lax Skin; Knee
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized to 2 treatment groups: "Right side treated" and "Left side treated". All subjects will receive three, single-sided injections of PLLA, performed 1 month apart. Treatments will be provided to one randomly assigned knee. The non-treatment knee will receive bacteriostatic water, injected in the same manner as PLLA. Up to one (1) syringe of PLLA, diluted at 16 mL, will be used per session
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Right Side Treated (Other): Subjects will be randomized to have their right side treated with PLLA and their left side treated with normal saline.
  Interventions: Device: poly-L-lactic acid to right knee
- Left Side Treated (Other): Subjects will be randomized to have their left side treated with PLLA and their right side treated with normal saline.
  Interventions: Device: poly-L-lactic acid to left knee

INTERVENTIONS:
Device: poly-L-lactic acid to right knee — Subjects will receive PLLA injections to the right knee and bacteriostatic water to the left.
  Other Names: Sculptra Aesthetic
  Arms: Right Side Treated
Device: poly-L-lactic acid to left knee — Subjects will receive PLLA injections to the left knee and bacteriostatic water to the right.
  Other Names: Sculptra Aesthetic
  Arms: Left Side Treated

SUMMARY:
All subjects will receive three, single-sided injections of PLLA, performed 1 month apart.

DETAILED DESCRIPTION:
Enrolled subjects will be randomized to 2 treatment groups: "Right side treated" and "Left side treated". All subjects will receive three, single-sided injections of PLLA, performed 1 month apart. Treatments will be provided to one randomly assigned knee. The non-treatment knee will receive bacteriostatic water, injected in the same manner as PLLA. Up to one (1) syringe of PLLA, diluted at 16 mL, will be used per session.

Subjects satisfying all inclusion and exclusion criteria will be enrolled in this trial. Prior to receiving any study treatment, mandatory photography using 2D photography and Vectra will be obtained of each subject's treatment area. All photographs may be used for research and/or commercial use.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women age 30 to 65 years of age.
2. Must be willing to give and sign an informed consent form and photographic release form.
3. Mild to Severe bilateral skin laxity above the knees (Upper Knee Laxity/Crepiness Grading Scale (Appendix B)
4. Must have had a stable body weight for at least 6 months prior to study entry.
5. Must be willing to maintain usual sun exposure, diet, and exercise routines for the duration of the study.
6. Negative urine pregnancy test results at the time of study entry (if applicable).
7. For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment participation.

   1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
   2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g. condoms and spermicide), abstinence and/or vasectomies of partner with a documented second acceptable method of birth control, should the subject become sexually active.
8. Must be willing to comply with study treatments and complete the entire course of the study.

Exclusion Criteria:

h. A subject with history of any other skin tightening procedures in the treatment area within the last 12 months. (Microfocused ultrasound, radiofrequency).

i. A subject with history of bio-stimulatory products or filler injections in the treatment area j. Subjects with scarring in treatment areas. k. A subject with tattoos or permanent implants in the treatment areas. l. A subject with history of or the presence of any skin condition/disease in the treatment area that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis).

m. A subject with an active bacterial, fungal, or viral infection in the treatment area.

n. A subject with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.

o. A subject planning any other cosmetic procedure to the study treatment area during the study period, other than the treatment that will be performed by the investigator.

p. Presence of incompletely healed wound in treatment area. q. Non-Ablative laser to the treatment area in the last 3 months. r. A female subject who is pregnant, nursing an infant or planning a pregnancy during the study.

s. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Investigator Assessed Improvement | Baseline to 6 Months post final treatment
  Blinded Investigator Grading

SECONDARY OUTCOMES:
Subject Assessed Improvement | Baseline to 6 Months post final treatment
  Subject Global Aesthetic Improvement Scale (SGIAS)
Subject Assessed Satisfaction | Baseline to 6 Months post final treatment
  Subject Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center, San Diego, California, United States